CLINICAL TRIAL: NCT01781169
Title: Health Effect of Oral Vitamin D Supplementation on Obese Chinese Males
Brief Title: Vitamin D Supplementation to Obese Chinese Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Center for Chronic Disease Control (Other)
Collaborators: Danone Institute China Diet Nutrition Research and Communication (Unknown)
Responsible Party: Principal Investigator, Zhou Ji-Chang, Vice Dean of Molecular Biology Lab, Shenzhen Center for Chronic Disease Control
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VD50kIU2011
Record Dates: First submitted 2013-01-25; First posted 2013-01-31 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Obesity; Insulin Resistance
Keywords: Vitamin D,; Oral supplementation,; Obese males
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obese group (Experimental): Oral supplementation of vitamin D (cholecalciferol), 50000 IU/wk for 8 weeks.
  Interventions: Dietary Supplement: Oral supplementation of vitamin D
- Normal-weight group (Experimental): Oral supplementation of vitamin D (cholecalciferol), 50000 IU/wk for 8 weeks.
  Interventions: Dietary Supplement: Oral supplementation of vitamin D

INTERVENTIONS:
Dietary Supplement: Oral supplementation of vitamin D — Weekly oral supplementation of 50,000 IU vitamin D (cholecalciferol) for eight weeks to the obese males compared with the normal-weight males. The chemical form of vitamin D is cholecalciferol capsuled as fine powder.

SUMMARY:
Hypothesis: Oral Supplementation of Vitamin D can Reduce Hypersecretion of Parathyroid Hormone and Insulin Resistance in Obese Chinese Males.

Protocol: Weekly oral supplementation of 50,000 IU vitamin D (cholecalciferol) or eight weeks to the obese males compared with the normal-weight males. Index measures were conducted at baseline and endpoint.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≥ 28kg/m2 or 18.5 ≤ BMI < 24 (kg/m2)
* non vegetarian Han Chinese and did not smoke, drink, nor take vitamin D supplements for > 2 y
* fasting serum glucose < 7.0 mmol/L
* serum glucose of 2 hr after 75 g oral glucose loading < 11.1 mmol/L
* normal functioning of liver and kidney evaluated by alkaline phosphatase, aspartate aminotransferase, creatinine, and uric acid

Exclusion Criteria:

* not match the above inclusion criteria
* diagnosed as having any organic diseases were excluded

Ages: 23 Years to 66 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Chang Zhou, Ph.D, Principal Investigator — Shenzhen Center for Chronic Disease Control
Locations (1):
- Shenzhen Center for Chronic Disease Control, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Heaney RP, Recker RR, Grote J, Horst RL, Armas LA. Vitamin D(3) is more potent than vitamin D(2) in humans. J Clin Endocrinol Metab. 2011 Mar;96(3):E447-52. doi: 10.1210/jc.2010-2230. Epub 2010 Dec 22. PMID 21177785
- [Result] Malabanan A, Veronikis IE, Holick MF. Redefining vitamin D insufficiency. Lancet. 1998 Mar 14;351(9105):805-6. doi: 10.1016/s0140-6736(05)78933-9. No abstract available. PMID 9519960
- [Result] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at a medical clinic (Health Service Center of Shuiku Community, Shenzhen, China) in May, 2011.
Pre-assignment Details: After enrollment, baseline information of the volunteers including vitamin D nutritional status, health records, etc. were evaluated. Including and excluding criteria were used to select the subjects who were suitable for the intervention trial.
Period: Overall Study
Arm/Group | Obese Group | Normal-weight Group
Started | 22 | 21
Completed | 21 | 21
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal-weight Group | Obese Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 34.4 (8) | 44.7 (8.8) | 39.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  China | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Plasma 25-hydroxy Vitamin D (25(OH)D) Level (Nmol/L)
Time Frame: Endpoint and baseline of the 8 weeks' trial
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Obese Group; Normal-weight Group: Oral supplementation of vitamin D.
Arm/Group | Obese Group | Normal-weight Group
Number analyzed (Participants) | 21 | 21
nmol/L
  Endpoint plasma 25(OH)D level | 116.7 (20.3) | 181.3 (30.2)
  Baseline plasma 25(OH)D level | 46.1 (9.1) | 52.8 (17.8)

ADVERSE EVENTS:
Time Frame: Eight weeks of the trial for all the participants.
Arm/Group | Normal-weight Group | Obese Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

LIMITATIONS AND CAVEATS:
The numbers of participants in both the obese group and normal-weight group were small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes